CLINICAL TRIAL: NCT01741415
Title: Distress Tolerance Treatment for Substance Users
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA032582 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2017-05

CONDITIONS: Substance Dependence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIDI (Experimental): Skills for Improving Distress Intolerance treatment protocol: individual, manualized treatment aimed at improving distress intolerance
  Interventions: Behavioral: SIDI
- SC (Placebo Comparator): supportive counseling; psychological placebo/talk therapy - aimed at controlling for non-specific therapeutic factors
  Interventions: Behavioral: SC

INTERVENTIONS:
Behavioral: SIDI
  Other Names: Skills for improving distress intolerance
  Arms: SIDI
Behavioral: SC
  Other Names: supportive counseling
  Arms: SC

SUMMARY:
Despite recent advances in substance abuse interventions, a large percentage of clients entering residential treatment for substance use will drop out of treatment prematurely, and of the remaining, many will relapse soon after treatment completion. Previous research indicates that an individual's ability to withstand psychological distress is a key factor necessary to maintain drug and alcohol abstinence and to remain in substance use treatment without absconding. In previous work, Dr. Bornovalova developed a specific distress tolerance treatment called Skills for Improving Distress Intolerance (SIDI). This intervention features skills training in behavioral and acceptance strategies and intentional clinical exposure to emotional distress. SIDI was developed and piloted with a sample of urban drug users seeking treatment in a residential facility. Individuals receiving SIDI exhibited greater improvement in distress tolerance than those in two comparison groups (receiving treatment-as-usual and supportive counseling).

Current study. The investigators received NIDA funding to conduct a randomized clinical trial with 325 clients entering a residential substance use treatment facility. Study participants will be randomized into two treatment groups: (1) those receiving SIDI and (2) those receiving Supportive Counseling (SC). Participants will receive 10 treatment sessions over a period of 4 months. Then, the investigators will follow clients for one year to examine treatment retention and abstinence.

ELIGIBILITY:
Inclusion criteria:

* 18-65 years of age
* Not evidencing severe cognitive deficits
* Ability to give informed consent

Exclusion criteria:

* <18 years of age or > 65 years of age
* Not evidencing severe cognitive deficits (site designation of 'not competent to stand trial')
* Unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2013-05-13; Primary Completion 2018-09-12 (Actual); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
abstinence at 1, 3, 6 & 12 month follow-up | 1, 3, 6 month follow-up post-treatment
  Measured via biological verification and timeline follow-back

SECONDARY OUTCOMES:
distress tolerance | 1, 3, 6 month follow-up
  ability to tolerate psychological distress

OTHER OUTCOMES:
successful/unsuccessful completion of residential addictions treatment | Baseline, post-treatment (at 3 month mark in residential facility), successful discharge within 6 months from residential facility
  successful/unsuccessful completion of residential addictions treatment
time in jail | 1, 3, 6 month follow-up in community
  measured by public records (# of days in jail by each timepoint)
psychiatric distress | post-treatment at 3 month mark in residential facility, 1, 3, 6 month follow-up in community
  psychiatric distress on brief symptom inventory
maladaptive personality | post-treatment (at 3 month mark in residential facility), 1, 3, 6 month follow-up in community
  change in maladaptive personality on the Personality Inventory for DSM5

CONTACTS AND LOCATIONS:
Locations (1):
- Agency for Community Treatment Services, Inc, Tarpon Springs, Florida, United States

REFERENCES:
- [Derived] Fatimah H, Hunter MD, Bornovalova MA. Modeling the dynamics of addiction relapse via the double-well potential system. J Psychopathol Clin Sci. 2025 Jan;134(1):69-80. doi: 10.1037/abn0000960. Epub 2024 Nov 14. PMID 39541537
- [Derived] Choate AM, Gorey C, Rappaport LM, Wiernik BM, Bornovalova MA. Alternative model of personality disorders traits predict residential addictions treatment completion. Drug Alcohol Depend. 2021 Nov 1;228:109011. doi: 10.1016/j.drugalcdep.2021.109011. Epub 2021 Sep 1. PMID 34521057